CLINICAL TRIAL: NCT07229612
Title: A Multicenter, Open-label Phase I/II Clinical Study on the Safety, Tolerability, Pharmacokinetics and Efficacy of SHR-4298 Injection in Patients With Malignant Solid Tumors
Brief Title: A Phase I/II Clinical Study of SHR-4298 Injection in Patients With Malignant Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-4298-101
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Malignant Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-4298 Group (Experimental)
  Interventions: Drug: SHR-4298 Injection

INTERVENTIONS:
Drug: SHR-4298 Injection — SHR-4298 injection.

SUMMARY:
This study is an open-label, multicenter Phase I/II clinical trial to evaluate the safety, tolerability and efficacy of SHR-4298 injection in patients with malignant solid tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must voluntarily agree to participate in the trial and sign a written informed consent form.
2. ECOG performance score of 0-1.
3. Life expectancy ≥ 3 months.
4. Have at least one measurable tumor lesion per RECIST v1.1.
5. Patients with recurrent or metastatic solid tumors confirmed by histopathology and not amenable to radical surgery or radical chemoradiotherapy.
6. Good level of organ function.
7. Provide archived or fresh tumor tissue for vendor test.

Exclusion Criteria:

1. Subjects with active central nervous system metastases or meningeal metastases.
2. Suffering from other malignant tumors within five years before the first use of the drug.
3. History of serious cardiovascular and cerebrovascular diseases.
4. Clinically significant bleeding symptoms occurred within 3 months before the first dose of study drug.
5. Subjects with uncontrolled tumor-related pain.
6. Clinically uncontrollable third space effusion or third space effusion requiring intervention within 7 days before the first study treatment.
7. Subjects who had a serious infection within 4 weeks before the first dose of the drug.
8. History of immunodeficiency, including a positive HIV test or active hepatitis B or C.
9. Subjects who received > 30 Gy of chest radiotherapy within 24 weeks before the first dose of the drug, subjects who received > 30 Gy of non-chest radiotherapy within 4 weeks before the first dose of the drug, and subjects who received ≤ 30 Gy of palliative radiation within 14 days before the first dose of the drug.
10. Underwent major organ surgery within 28 days before the first dose of the drug.
11. Those who are known to be allergic to any ingredients or excipients of SHR-4298 product.
12. Administered a live attenuated vaccine within 28 days before the first dose.
13. Female subjects who are pregnant, breastfeeding, or planning to become pregnant during the study.
14. Per the investigator's judgment, there are any other circumstances that may increase the risk of participating in the study, interfere with the study results, or make participation in the study inappropriate.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs). | Approximately 18 months.
Incidence and severity of serious adverse events (SAEs). | Approximately 18 months.
Maximum Tolerated Dose (MTD). | Approximately 18 months.
Maximum Applicable Dose (MAD). | Approximately 18 months.
Recommended Phase 2 Dose (RP2D). | Approximately 18 months.
Dose-limiting toxicity (DLT). | Approximately 18 months.

SECONDARY OUTCOMES:
Overall response rate (ORR). | Approximately 18 months.
Duration of response (DoR). | Approximately 18 months.
Disease control rate (DCR). | Approximately 18 months.
Progression-free survival (PFS). | Approximately 18 months.
Overall survival (OS). | Approximately 5 years after the last subject enrolled.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided